CLINICAL TRIAL: NCT01932762
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of a Combination Regimen of MK-5172 With/Without MK-8742 and/or Ribavirin (RBV) in Treatment-naive Subjects With Chronic Hepatitis C Genotype 2, 4, 5 and 6 Infection
Brief Title: Efficacy and Safety of Combination Grazoprevir (MK-5172) + Elbasvir (MK-8742) + Ribavirin (RBV) in Genotype 2 Hepatitis C Infection (MK-5172-047)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-047; 2013-002169-21 (EudraCT Number)
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GT2: Grazoprevir + Elbasvir + RBV (Arm A1) (Experimental): During Part A of the study, GT2 participants will receive 100 mg grazoprevir + 50 mg elbasvir + standard weight-based dosing of RBV for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- GT2: Grazoprevir + RBV (Arm B1) (Experimental): During Part B of the study, GT2 participants will receive 100 mg grazoprevir + standard weight-based dosing of RBV for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Ribavirin
- GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) (Experimental): During Part B of the study, GT4/GT5/GT6 participants will receive 100 mg grazoprevir + 50 mg elbasvir + standard weight-based dosing of RBV for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- GT 4,5,6: Grazoprevir + Elbasvir (Arm B3) (Experimental): During Part B of the study, GT4/GT5/GT6 participants will receive 100 mg grazoprevir + 50 mg elbasvir for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir

INTERVENTIONS:
Drug: Grazoprevir — 100 mg every day (QD) orally
  Other Names: MK-5172
Drug: Elbasvir — 50 mg QD orally
  Other Names: MK-8742
  Arms: GT 4,5,6: Grazoprevir + Elbasvir (Arm B3); GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2); GT2: Grazoprevir + Elbasvir + RBV (Arm A1)
Drug: Ribavirin — Administered twice daily (BID) orally at a total daily dose of 800 mg to 1400 mg based on participant's weight on Day 1
  Other Names: Rebetol™
  Arms: GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2); GT2: Grazoprevir + Elbasvir + RBV (Arm A1); GT2: Grazoprevir + RBV (Arm B1)

SUMMARY:
This is a multi-site, open-label trial evaluating the safety and efficacy of 100 mg of grazoprevir (MK-5172) used in combination with or without 50 mg of elbasvir (MK-8742) and/or ribavirin (RBV) in treating non-cirrhotic treatment-naïve participants with chronic genotype (GT) 2, 4, 5, and 6 hepatitis C infection.

In Part A there is no randomization or stratification; all GT2 participants will be assigned to arm A1. In Part B, all GT2 participants will be assigned to Arm B1 and all participants with GT4, GT5 and GT6 will be randomized in a 1:1 ratio to either Arm 3 or Arm 4 with stratification by genotype.

ELIGIBILITY:
Inclusion Criteria:

Parts A and B: -Body weight ≥50 kg (111 lbs) and ≤ 125 kg (275 lbs) -Has absence of cirrhosis -Agrees to use two acceptable methods of birth control from at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study drug, or longer if dictated by local regulations (for female participant who is of childbearing potential or male participant with female sexual partner who is of childbearing potential).

Part A only: -Has chronic HCV GT2 infection Part B only: -Has chronic HCV GT2, GT4, GT5, or GT6 infection

Exclusion Criteria:

Parts A and B:

-Is not treatment naïve (participant has had previous treatment with any interferon, RBV, approved or experimental direct acting antiviral(s), or other investigational therapies for HCV) -Is determined to be coinfected with hepatitis B virus (HBsAg positive) or HIV -Has evidence of, or is under evaluation for, hepatocellular carcinoma (HCC) -Has a clinical diagnosis of substance abuse including the following specified drugs within specified timeframes: Alcohol, intravenous drugs, inhalational, psychotropics, narcotics, cocaine use, prescription or over-the-counter drugs (within 1 year of the screening visit), is receiving opiate agonist substitution therapy (within 1 year of screening visit), or excessive historic marijuana use -Has evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years -Female participant who is pregnant, lactating, expecting to conceive or donate eggs, or is of childbearing potential and unwilling to commit to two methods of birth control throughout treatment and after the completion of all treatment, or male participant who is planning to impregnate or provide sperm donation or has a female sexual partner of childbearing potential and is unwilling to commit to using a two methods of birth control throughout treatment and after the completion of all treatment -Has evidence or history of chronic hepatitis not caused by HCV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, and autoimmune hepatitis. -Has uncontrolled diabetes (documented HbA1c >8.5%)

Part A only:

-Has non GT2 HCV infection

Part B only:

-Has HCV infection with a genotype other than GT2, GT4, GT5 or GT6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-12-04 (Actual); Study Completion 2014-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Brown A, Hezode C, Zuckerman E, Foster GR, Zekry A, Roberts SK, Lahser F, Durkan C, Badshah C, Zhang B, Robertson M, Wahl J, Barr E, Haber B; C-SCAPE Study Investigators. Efficacy and safety of 12 weeks of elbasvir +/- grazoprevir +/- ribavirin in participants with hepatitis C virus genotype 2, 4, 5 or 6 infection: The C-SCAPE study. J Viral Hepat. 2018 May;25(5):457-464. doi: 10.1111/jvh.12801. Epub 2018 Mar 14. PMID 29152828
- [Derived] Asselah T, Reesink H, Gerstoft J, de Ledinghen V, Pockros PJ, Robertson M, Hwang P, Asante-Appiah E, Wahl J, Nguyen BY, Barr E, Talwani R, Serfaty L. Efficacy of elbasvir and grazoprevir in participants with hepatitis C virus genotype 4 infection: A pooled analysis. Liver Int. 2018 Sep;38(9):1583-1591. doi: 10.1111/liv.13727. Epub 2018 Mar 31. PMID 29461687

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 98 participants were assigned to treatment at 28 sites worldwide and all enrolled participants received ≥1 dose of study therapy. 30 participants enrolled in Part A and 68 were enrolled and randomized in Part B of the study. Enrollment in Part C, an evaluation of a fixed-dose combination of grazoprevir and elbasvir, was never initiated.
Groups:
- GT2: Grazoprevir + Elbasvir + RBV (Arm A1): During Part A of the study, GT2 participants received 100 mg grazoprevir plus 50 mg elbasvir plus standard weight-based dosing of ribavirin (RBV) for 12 weeks.
- GT2: Grazoprevir + RBV (Arm B1): During Part B of the study, GT2 participants received 100 mg grazoprevir plus standard weight-based dosing of RBV for 12 weeks.
- GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2): During Part B of the study, GT4/GT5/GT6 participants received 100 mg grazoprevir plus 50 mg elbasvir plus standard weight-based dosing of RBV for 12 weeks.
- GT 4,5,6: Grazoprevir + Elbasvir (Arm B3): During Part B of the study, GT4/GT5/GT6 participants received 100 mg grazoprevir plus 50 mg elbasvir for 12 weeks.
Period: Overall Study
Arm/Group | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) | GT2: Grazoprevir + RBV (Arm B1) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3)
Started | 30 | 30 | 19 | 19
Completed | 24 | 28 | 19 | 18
Not Completed | 6 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GT2: Grazoprevir + Elbasvir + RBV (Arm A1): During Part A of the study, GT2 participants received 100 mg grazoprevir plus 50 mg elbasvir plus standard weight-based dosing of RBV for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) | GT2: Grazoprevir + RBV (Arm B1) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3) | Total
Number analyzed (Participants) | 30 | 30 | 19 | 19 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (13.6) | 48.3 (14.6) | 52.2 (9.3) | 52.8 (12.3) | 49.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 11 | 7 | 42
  Male | 19 | 17 | 8 | 12 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After The End of Study Therapy (SVR12)
Description: SVR12 was defined as Hepatitis C Virus ribonucleic acid (HCV RNA) <25 IU/mL, either target detected but unquantifiable (TD[u]) or target not detected (TND), at 12 weeks after the end of all study therapy. The percentage of participants with SVR12 and accompanying 95% confidence intervals (CIs) were reported for each treatment arm in the Per-Protocol (PP) Population.
Time Frame: 12 weeks after end of all therapy (Study Week 24)
Population: All participants in the PP Population (all randomized participants receiving ≥1 dose of study therapy with no important protocol deviations) with available data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) | GT2: Grazoprevir + RBV (Arm B1) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3)
Number analyzed (Participants) | 27 | 24 | 17 | 13
percentage of participants | 85.2 [66.3 to 95.8] | 75.0 [53.3 to 90.2] | 94.1 [71.3 to 99.9] | 76.9 [46.2 to 95.0]

2. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Serious AEs (SAEs), Drug-Related AEs, Drug-Related SAEs, or Discontinuation of Study Treatment Due to AE During the Treatment Period and First 14 Follow-up Days
Description: AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. An SAE was an AE that resulted in death, was life threatening, resulted in persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a cancer, was associated with an overdose, was another important medical event. The investigator determined the relationship of the AE to the treatment as unrelated or possibly, probably, or definitely related.
Time Frame: Treatment period plus the first 14 days of follow-up (up to 14 weeks)
Population: All-Subjects-As-Treated (ASAT) Population; all randomized participants who received ≥ 1 dose of study therapy. The percentage of participants with specific AEs and accompanying 95% CI were reported for each treatment arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) | GT2: Grazoprevir + RBV (Arm B1) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3)
Number analyzed (Participants) | 30 | 30 | 19 | 19
percentage of participants
  AEs | 86.7 [69.3 to 96.2] | 86.7 [69.3 to 96.2] | 94.7 [74.0 to 99.9] | 78.9 [54.4 to 93.9]
  SAEs | 3.3 [0.1 to 17.2] | 3.3 [0.1 to 17.2] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 17.6]
  Drug-related AE | 63.3 [43.9 to 80.1] | 63.3 [43.9 to 80.1] | 57.9 [33.5 to 79.7] | 36.8 [16.3 to 61.6]
  Drug-related SAE | 0.0 [0.0 to 11.6] | 3.3 [0.1 to 17.2] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 17.6]
  Discontinuation due to AE | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 17.6] | 5.3 [0.1 to 26.0]

3. Secondary Outcome: Mean Time to First Achievement of Undetectable HCV RNA During Treatment
Description: HCV-RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test (v.2.0) on blood samples drawn from each participant during treatment at TWs 1, 2, 4, 8, and 12. Undetectable HCV RNA (or TND) was defined as below the 9.3 IU/ml limit of detection. Kaplan Meier summary statistics were calculated for each treatment arm in the Full Analysis Set (FAS).
Time Frame: From TW1 until first achievement of undetectable HCV RNA (up to 12 weeks)
Population: FAS; all randomized participants who received ≥1 dose of study therapy. Participants in the FAS not achieving TND were censored from the analysis.
Measure: Mean (Standard Error); unit: days
Arm/Group | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) | GT2: Grazoprevir + RBV (Arm B1) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3)
Number analyzed (Participants) | 30 | 26 | 19 | 18
days | 25.2 (2.8) | 26.9 (3.0) | 27.4 (4.5) | 21.3 (1.7)

4. Secondary Outcome: Percentage of Participants Achieving Undetectable HCV RNA During Treatment By Timepoint
Description: HCV-RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test (v.2.0) on blood samples drawn from each participant during treatment at TWs 1, 2, 4, 8, and 12. Undetectable HCV RNA (or TND) was defined as below the 9.3 IU/ml limit of detection. The percentage of participants achieving undetectable HCV RNA and accompanying 95% CIs were reported at TW2, TW4, and TW12 for each treatment arm of the PP Population.
Time Frame: From TW 2 through TW 12 (up to 12 weeks)
Population: All participants in the PP Population (all randomized participants receiving ≥1 dose of study therapy and with no important protocol deviations) with available data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) | GT2: Grazoprevir + RBV (Arm B1) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3)
Number analyzed (Participants) | 28 | 24 | 17 | 15
percentage of participants
  Week 2 (n=28, 24, 16, 15) | 42.9 [24.5 to 62.8] | 50.0 [29.1 to 70.9] | 50.0 [24.7 to 75.3] | 53.3 [26.6 to 78.7]
  Week 4 (n=28, 24, 17, 15) | 85.7 [67.3 to 96.0] | 79.2 [57.8 to 92.9] | 88.2 [63.6 to 98.5] | 80.0 [51.9 to 95.7]
  Week 12 (n=28, 24, 17, 14) | 96.4 [81.7 to 99.9] | 83.3 [62.6 to 95.3] | 100.0 [80.5 to 100.0] | 78.6 [49.2 to 95.3]

5. Secondary Outcome: Percentage of Participants Achieving HCV RNA <25 IU/mL During Treatment By Timepoint
Description: HCV-RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test (v.2.0) on blood samples drawn from each participant during treatment at TWs 1, 2, 4, 8, and 12. The Roche COBAS™ Taqman™ HCV Test (v.2.0) has a lower limit of quantification (LLoQ) of 25 IU/ml and a limit of detection of 9.3 IU/ml. The percentage of participants with HCV RNA levels <25 IU/ml (either TD[u] or TND) and accompanying 95% CIs were reported at TW2, TW4, and TW12 for each treatment arm of the PP Population.
Time Frame: From TW 2 through TW 12 (up to 12 weeks)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) | GT2: Grazoprevir + RBV (Arm B1) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3)
Number analyzed (Participants) | 28 | 24 | 17 | 15
percentage of participants
  Week 2 (n=28, 24, 16, 15) | 96.4 [81.7 to 99.9] | 79.2 [57.8 to 92.9] | 87.5 [61.7 to 98.4] | 93.3 [68.1 to 99.8]
  Week 4 (n=28, 24, 17, 15) | 100.0 [87.7 to 100.0] | 91.7 [73.0 to 99.0] | 100.0 [80.5 to 100.0] | 93.3 [68.1 to 99.8]
  Week 12 (n=28, 24, 17, 14) | 96.4 [81.7 to 99.9] | 87.5 [67.6 to 97.3] | 100.0 [80.5 to 100.0] | 85.7 [57.2 to 98.2]

6. Secondary Outcome: Percentage of Participants Achieving SVR4
Description: SVR4 was defined as HCV RNA <25 IU/mL, either TD(u) or TND, at 4 weeks after the end of all study therapy. The percentage of participants with SVR4 and accompanying 95% CIs were reported for each treatment arm of the PP Population.
Time Frame: 4 weeks after end of all therapy (Study Week 16)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) | GT2: Grazoprevir + RBV (Arm B1) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3)
Number analyzed (Participants) | 27 | 24 | 17 | 14
percentage of participants | 88.9 [70.8 to 97.6] | 83.3 [62.6 to 95.3] | 94.1 [71.3 to 99.9] | 78.6 [49.2 to 95.3]

7. Secondary Outcome: Percentage of Participants Achieving SVR24
Description: SVR24 was defined as HCV RNA <25 IU/mL, either TD(u) or TND, at 24 weeks after the end of all study therapy. The percentage of participants with SVR24 and accompanying 95% CIs were reported for each treatment arm of the PP Population.
Time Frame: 24 weeks after end of all therapy (Study Week 36)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) | GT2: Grazoprevir + RBV (Arm B1) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3)
Number analyzed (Participants) | 26 | 24 | 17 | 13
percentage of participants | 84.6 [65.1 to 95.6] | 75.0 [53.3 to 90.2] | 94.1 [71.3 to 99.9] | 76.9 [46.2 to 95.0]

ADVERSE EVENTS:
Time Frame: From TW1 through FW 24 (up to 36 weeks)
Description: AEs were reported for the ASAT Population (all randomized participants who received ≥1 dose of study therapy) for both the treatment and follow-up periods.
Arm/Group | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) | GT2: Grazoprevir + RBV (Arm B1) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3)
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/30 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 26/30 | 25/30 | 18/19 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) (N=30) | GT2: Grazoprevir + RBV (Arm B1) (N=30) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) (N=19) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3) (N=19)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GT2: Grazoprevir + Elbasvir + RBV (Arm A1) (N=30) | GT2: Grazoprevir + RBV (Arm B1) (N=30) | GT 4,5,6: Grazoprevir + Elbasvir + RBV (Arm B2) (N=19) | GT 4,5,6: Grazoprevir + Elbasvir (Arm B3) (N=19)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces pale (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (6) | 2 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 5 (6) | 2 (3) | 0 (0) | 1 (1)
Asthenia (General disorders) | 5 (5) | 6 (6) | 3 (3) | 4 (4)
Chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 12 (13) | 6 (7) | 5 (5) | 3 (3)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Thirst (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 4 (7) | 4 (6) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inflammation of wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 1 (1) | 3 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 1 (2) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 4 (5) | 6 (8) | 5 (20)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 1 (1) | 3 (3) | 2 (3)
Irritability (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital tract inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 4 (4) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 2 (3) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 3 (5) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.